CLINICAL TRIAL: NCT07158281
Title: Investigation of the Effects of Dual-Tasking on Gait Variability and Symmetry in Individuals With Nonspecific Neck Pain
Brief Title: Dual-Task Effects on Gait in Nonspecific Neck Pain
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Güngör Beyza ÖZVAR, Principal Investıgator, Hacettepe University
Other Study IDs: non-spesific neck pain
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Neck Pain; Gait
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nonspecific Neck Pain: Adults aged 18-60 with chronic nonspecific neck pain (≥3 months), scoring ≥10 on the Neck Disability Index, no neurological/systemic disease, no prior cervical surgery.
- Healthy Control: Age- and sex-matched adults without neck pain or neurological/systemic disorders.

SUMMARY:
The aim of this study is to examine the impact of motor and cognitive dual-task conditions on gait variability and gait symmetry in individuals with NSNP, compared with healthy controls. This cross-sectional trial will recruit participants aged 18-60, including 21 patients with NSNP and 21 age-matched healthy controls. Gait parameters will be assessed using a wearable sensor system (BTS G-Walk). Primary outcomes are gait variability and gait symmetry under single-task, motor dual-task, and cognitive dual-task walking conditions.

DETAILED DESCRIPTION:
Each participant will complete three walking conditions:

Single-task walking (walking at a self-selected pace), Motor dual-task walking (walking while carrying a tray with a glass of water), and Cognitive dual-task walking (walking while verbally reporting the number of letters in presented words).

Gait parameters will be measured using the BTS G-Walk wearable sensor system, which records accelerometric data at the lumbar level (L4-L5) and calculates temporospatial parameters. Gait variability will be quantified using the coefficient of variation formula, and gait symmetry will be determined using symmetry index calculations.

The primary outcomes are gait variability and gait symmetry across the three walking conditions. Secondary outcomes include pain characteristics, the Neck Disability Index (NDI), and the Bournemouth Neck Questionnaire (BNQ).

The study hypothesizes that both motor and cognitive dual-task conditions will significantly affect gait variability and symmetry in individuals with NSNP, and these effects will differ from those observed in healthy controls. Findings are expected to improve understanding of motor control alterations in NSNP and provide guidance for individualized rehabilitation programs and therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* for NSNP group:

  * Adults aged 18-60 years
  * History of nonspecific neck pain lasting at least 3 months
  * Neck Disability Index (NDI) score ≥10
  * Willingness to participate and provide informed consent
* for the Healthy Control group

  * Adults aged 18-60 years
  * No history of neck pain or musculoskeletal/neurological/systemic disorders
  * Willingness to participate and provide informed consent

Exclusion Criteria:(applies to both groups):

* Previous spinal surgery
* History of traumatic cervical injury
* Diagnosed cervical radiculopathy, spondylosis, spondylolisthesis, or disc herniation
* Presence of any neurological or systemic disease
* Musculoskeletal disorders affecting gait performance
* Cognitive impairment or psychiatric conditions interfering with test participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of adults aged 18-60 years, including individuals with chronic nonspecific neck pain (NSNP) and age-matched healthy volunteers. Participants will be recruited from the students, staff, and first-degree relatives of Yüksek İhtisas University, Faculty of Health Sciences.
  The NSNP group will include participants with a history of neck pain lasting at least three months and a Neck Disability Index (NDI) score of ≥10. The control group will include individuals without neck pain or neurological, systemic, or musculoskeletal disorders.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Gait Variability | up to 3 months
  Gait variability calculated using the coefficient of variation.Gait variability is the ratio of the mean to the standard deviation and is calculated as a percentage. The score ranges from 0 to 100. A higher score indicates greater variability and decreased gait control. formula.
  Measurement Tool: BTS G-Walk wearable sensor system.
Gait Symmetry | up to 3 months
  Symmetry Index (SI) of spatiotemporal gait parameters between right and left limbs, calculated with the standard formula.Measurement Tool: BTS G-Walk wearable sensor system.Gait symmetry is calculated using a formula that compares the right and left extremities. "0" indicates complete symmetry, while "≥1" indicates asymmetry.
Pain Intensity | Assessed at baseline.
  Neck pain intensity measured using the Visual Analog Scale (VAS, 0-10).
Neck Disability Index (NDI) | Assessed at baseline (only in NSNP group).
  Self-reported questionnaire assessing functional disability related to neck pain. Validated Turkish version will be used.he NDI is a 10-item questionnaire assessing neck pain-related disability in daily life (e.g., pain intensity, personal care, concentration, work, driving, sleeping).Each item is scored from 0 to 5 (0 = no disability, 5 = maximum disability). The total score ranges from 0 to 50.
Bournemouth Neck Questionnaire (BNQ) | Assessed at baseline (only in NSNP group).
  elf-reported questionnaire evaluating pain severity, emotional distress, fear of movement, and coping strategies. Validated Turkish version will be used.The BNQ is a 7-item questionnaire evaluating the impact of neck pain on pain severity, activities of daily living, emotional well-being, anxiety/depression, fear of movement (kinesiophobia), and coping strategies.
  Scoring: Each item is scored on a 0-10 numeric rating scale (0 = no problem, 10 = maximum problem). The total score ranges from 0 to 70.
  Interpretation: Higher scores indicate greater disability and psychosocial impact of neck pain.

CONTACTS AND LOCATIONS:
Overall Officials: Busra Kalkan Balak, Principal Investigator — Yuksek Ihtisas University; Elıf Sena Colak, Principal Investigator — Yuksek Ihtisas University; Aslı Isıkdemır, Principal Investigator — Yuksek Ihtisas University; Demet Cıhan, Principal Investigator — Yuksek Ihtisas University
Locations (1):
- Yuksek Ihtisas University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No